CLINICAL TRIAL: NCT03133273
Title: Study of the Therapeutic Response and Survival of Patients with Metastatic Colorectal Cancer (stage IV) and Treated According to the Guidelines of a Chemosensitivity Test, Oncogramme®
Brief Title: Study of the Therapeutic Response and Survival of Patients with Metastatic Colorectal Cancer (stage IV) and Treated According to the Guidelines of a Chemosensitivity Test, Oncogramme® (ONCOGRAM)
Acronym: ONCOGRAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Oncomédics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: I16014 (ONCOGRAM)
Record Dates: First submitted 2017-04-20; First posted 2017-04-28 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer Metastatic; Chemotherapy
Keywords: Colorectal Cancer Metastatic; Chemosensitivity

STUDY DESIGN:
Intervention Model Description: Patients corresponding to the inclusion criteria and having a histologically proven metastatic CRC on biopsies or primary tumor excision and / or one or more metastatic sites will be recruited prospectively and randomized into two groups.
  1. Usual care group: no Oncogramme will be made.
  2. Oncogramme group: Taking of tumor fragments on the histological piece by an anatomopathological physician at the time of the histological examination and placing samples in the transport medium. The Oncogramme will be performed by Oncomedics on all specimens. Results will be returned to clinicians within 15 days.
  For both groups, the adjuvant treatment will be decided in the multidisciplinary consultation meeting (MCM), according to the recommendations in force and adapted to the general medical condition of the patient. For patients in the Oncogramme group, chemotherapy will be adapted to Oncogramme.
Who Masked: Participant
Masking Description: The result of Oncogramme® will not give to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Patient is followed within the usual care for stage 4 colorectal cancer
- Oncogramme® (Experimental): For patients in the Oncogramme® group, chemotherapy will be adapted to Oncogramme® results.
  Interventions: Other: Oncogramme®

INTERVENTIONS:
Other: Oncogramme® — Patient is followed within the usual care for stage 4 colorectal cancer, but an Oncogramme test will be made and chemotherapy will be adapted to the results.
  Arms: Oncogramme®

SUMMARY:
Currently, chemotherapies are empirically administered to patients treated for colorectal cancer (CRC). Selection is based on the efficacy of a protocol previously determined on the largest number (consensus treatment), the decision-making process being weighted by patient's intrinsic criteria. However, each patient is unique, due to the inter- and intratumoral heterogeneity inherent in any cancer, partly explaining the unsatisfactory response rates observed for available chemotherapies. Functional sensitivity tests offer the possibility to adapt the treatment to each patient: they are based on an ex vivo study of the responses of the tumor cells (survival / death) to the different molecules / therapeutic combinations (chemotherapy or targeted therapy) likely to be administered to the patient. This response, translated into a tumor-specific sensitivity profile, can be used by the clinicians to determine the most appropriate therapeutic protocol. By increasing the therapeutic efficacy from the first line and reducing the deleterious side effects associated with multiple drug cycles, the sensitivity test transforms the consensus approach into personalized medicine, providing patients with improved progression free survival (PFS) associated with an improvement in the quality of life. Oncomedics has developed Oncogramme®, a CE-labeled in vitro diagnostic medical device that has already demonstrated the ability to predict chemosensitivity in a recent pilot study of metastatic CRC (prediction with 84% chance of success of tumor sensitivity to chemotherapy, vs. 50% maximum for chemotherapy administered according to the consensus method). The hypothesis that patients treated with a metastatic CRC for which systemic chemotherapy is adapted using Oncogramme® have better response rates, PFS and quality of life than patients treated according to usual practice, with optimization of the costs of care. To our knowledge, this is the only fully standardized test available, where each step and reagents of the procedure are mastered. The reliability of the procedure makes it possible to render a personalized result for each patient in 97% of the cases. In addition, the analysis is specifically centered on tumor cells using a method using fully defined, developed and validated media and reagents for each cancer, including CRC. The method of revealing the effect of the therapies identifies the proportion of dead cells in each condition, whatever their physiological state (proliferation / quiescence), by determining the percentage of living and killed cells, thus ensuring high sensitivity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with metastatic colon or rectal adenocarcinoma (Stage IV) who can benefit from standard systemic chemotherapy (monotherapy based on 5-FU, polychemotherapy type FOLFOX, FOLFIRI, FOLFIRINOX, associated or not with targeted therapies Adapted to the expression of BRAF and RAS, whatever the route of administration of the proposed, oral or intravenous therapies)
* Metastatic CRC diagnosed preoperatively on imaging or per-operative on macroscopic findings and proved by histological analysis (biopsy or surgical excision and if possible biopsies or excrescence on the metastatic sites)
* Measurable metastases according to RECIST
* Chemotherapy for curative or palliative purposes
* Patient with consent.
* Affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* Formal contraindication to paraclinic exploration essential for patient follow-up
* Exclusive use of radiotherapy, targeted therapy, immunotherapy or hormone therapy, exclusive palliative support
* Patient with an absolute contraindication to the administration of chemotherapy
* Pregnant, lactating or non-contraceptive women for childbearing age women
* Patient with a difficulty of understanding the protocol
* Patient under protective measures (guardianship, curatorship, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of the progression or death of the patient. | Year 1
  The event studied is the occurrence of the progression or death of the patient during the year following the inclusion in the study. The progression of the patient is determined by the RECIST (Response Evaluation Criteria in Solid Tumors).

SECONDARY OUTCOMES:
Response to first-line treatment administrated | every month, up to 12 months
  Percentage of patients in each response category to first-line treatment administered, evaluated by RECIST in each of the two groups.
Overall survival | Month 6 and Year 1
  The event study is the death of the patient during the 6 months and the year following the inclusion.
Specific survival | Month 6 and Year 1
  The event considered is death due to illness during the 6 months and the year following the inclusion. The attribution of the death to the illness will be made by the adjudication committee.
Incremental Cost / Efficiency Ratio | Year 1
  Calculation of the Incremental Cost / Efficiency Ratio (ICER) expressed in euros per year of life gained without occurrence of death or progression to 1 year of the adapted chemotherapeutic treatment according to the results of Oncogramme® using EQ5D-5L s
Incremental Cost / Utility Ratio | Year 1
  Calculation of the Incremental Cost / Utility Ratio (ICUR) expressed in euros per QALY gained at 1 year of the adapted chemotherapeutic treatment according to the results of Oncogramme® using EQ5D-5L scale.
Quality of life | Month 3, Month 6, Month 9 and Year 1
  Compare the quality of life of patients at 3 months, 6 months, 9 months and 1 year between the two groups using the EQ5D-5L questionary score.
No adaptation of chemotherapy | every month, up to 12 months
  If there is no adaptation of the treatment to the results of Oncogramme®, describe the criteria that led to the failure to take into account the results of Oncogramme®
Grade 3 and higher adverse events related to chemotherapy | Year 1
  Describe and compare in both groups the proportion of grade 3 and higher adverse events related to chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Mathonnet, MD, Principal Investigator — University Hospital, Limoges
Locations (13):
- France (13):
  - CHU d'AMIENS, Amiens
  - Bergonié Institut, Bordeaux
  - Clinique des Cédres, Brive-la-Gaillarde
  - CHU de TOURS, Chambray-lès-Tours
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - CHu de la Martinique, Fort-De-France
  - Hospital Center, Guéret
  - Limoges University Hospital, Limoges
  - Nimes University Hospital, Nîmes
  - CHU de POITIERS, Poitiers
  - CH de Saint Junien, Saint-Junien
  - Centre Médical MGEN Alfred Leune, Sainte-Feyre
  - CHU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathonnet M, Vanderstraete M, Bounaix Morand du Puch C, Giraud S, Lautrette C, Ouaissi M, Tabchouri N, Taibi A, Martin R, Herafa I, Tchalla A, Christou N; ONCOGRAM trial investigators. ONCOGRAM: study protocol for the evaluation of therapeutic response and survival of metastatic colorectal cancer patients treated according to the guidelines of a chemosensitivity assay, the Oncogramme(R). Trials. 2021 Aug 21;22(1):556. doi: 10.1186/s13063-021-05531-y. PMID 34419125